CLINICAL TRIAL: NCT04908202
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Deucravacitinib in Participants With Active Psoriatic Arthritis Who Are Naïve to Biologic Disease-modifying Anti-rheumatic Drugs
Brief Title: A Study to Determine the Efficacy and Safety of Deucravacitinib Compared With Placebo in Participants With Active Psoriatic Arthritis (PsA) Who Are Naïve to Biologic Disease-modifying Anti-rheumatic Drugs
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM011-054; 2023-506256-25 (Other: EU Trial Number); U1111-1259-9443 (Registry Identifier: WHO)
Record Dates: First submitted 2021-05-28; First posted 2021-06-01 (Actual); Results first posted 2025-10-24 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Psoriatic Arthritis
Keywords: Biologic-Naive; BMS-986165; Deucravacitinib; Disease-modifying Anti-rheumatic Drugs; DMARDs; Joint Disease; Psoriatic Arthritis; PsA
MeSH Terms: conditions — Arthritis, Psoriatic; Joint Diseases | interventions — deucravacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Deucravacitinib (Experimental)
  Interventions: Drug: Deucravacitinib
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Deucravacitinib — Specified dose on specified days
  Other Names: BMS-986165
  Arms: Deucravacitinib
Other: Placebo — Specified dose on specified days
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of deucravacitinib versus placebo in participants with active psoriatic arthritis who are naïve to biologic disease-modifying anti-rheumatic drugs. The long term extension period will provide additional long-term efficacy and safety information.

ELIGIBILITY:
Inclusion Criteria

* Diagnosed to have psoriatic arthritis (PsA) of at least 3 months duration at screening.
* Meets the Classification Criteria for Psoriatic Arthritis at Screening.
* Active plaque psoriatic skin lesion(s) or documented medical history of plaque psoriasis (PsO) at screening.
* Active arthritis as shown by ≥ 3 swollen joints and ≥ 3 tender joints at Screening and day 1.
* Participant has high sensitivity C-reactive protein (hsCRP) ≥ 3 mg/L at Screening.
* ≥ 1 PsA-related hand and/or foot joint erosion on X-ray during Screening Period that is confirmed by central reading.
* Must have completed the week 52 treatment for the optional open-label long-term extension period.

Exclusion Criteria

* Nonplaque psoriasis at screening or day 1.
* Other autoimmune condition such as systemic lupus erythematous, mixed connective tissue disease, multiple sclerosis, or vasculitis.
* History of or current inflammatory joint disease other than PsA (e.g., gout, reactive arthritis, rheumatoid arthritis, ankylosing spondylitis, Lyme disease).
* Active fibromyalgia.
* Received an approved or investigational biologic therapy for the treatment of PsA or PsO.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 670 (Actual)
Dates: Start 2021-07-13 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2027-06-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (183):
- United States (33):
  - Local Institution - 0197, Gilbert, Arizona
  - Local Institution - 0188, Jonesboro, Arkansas
  - Local Institution - 0168, Fontana, California
  - Local Institution - 0199, Fullerton, California
  - Local Institution - 0038, Sacramento, California
  - Cohen Medical Centers, Thousand Oaks, California
  - Local Institution - 0170, Denver, Colorado
  - Local Institution - 0195, Clearwater, Florida
  - Local Institution - 0272, Margate, Florida
  - Local Institution - 0082, Miami Lakes, Florida
  - Local Institution - 0171, Gainesville, Georgia
  - Local Institution - 0087, Boise, Idaho
  - Local Institution - 0080, Chicago, Illinois
  - Local Institution - 0177, Orland Park, Illinois
  - Local Institution - 0178, Schaumburg, Illinois
  - Local Institution - 0083, Lexington, Kentucky
  - Local Institution - 0042, Hagerstown, Maryland
  - Local Institution - 0198, Detroit, Michigan
  - Local Institution - 0201, Springfield, Missouri
  - Local Institution - 0268, Kalispell, Montana
  - Local Institution - 0186, Voorhees Township, New Jersey
  - University Hospitals Cleveland Medical Center-Dermatology, Cleveland, Ohio
  - Local Institution - 0028, Middleburg Heights, Ohio
  - Local Institution - 0179, Perrysburg, Ohio
  - Local Institution - 0182, Oklahoma City, Oklahoma
  - Local Institution - 0185, Corvallis, Oregon
  - Local Institution - 0175, Greenville, South Carolina
  - Local Institution - 0036, Jackson, Tennessee
  - Local Institution - 0172, Allen, Texas
  - Local Institution - 0189, Amarillo, Texas
  - Local Institution - 0032, Dallas, Texas
  - Local Institution - 0273, Bothell, Washington
  - Local Institution - 0181, Beckley, West Virginia
- Argentina (10):
  - Local Institution - 0213, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Local Institution - 0054, La Plata, Buenos Aires
  - Local Institution - 0215, Quilmes, Buenos Aires
  - Local Institution - 0046, Córdoba, Córdoba Province
  - Local Institution - 0196, Rosario, Santa Fe Province
  - Local Institution - 0047, San Miguel de Tucumán, Tucumán Province
  - Local Institution - 0194, Buenos Aires
  - Local Institution - 0169, Buenos Aires
  - Local Institution - 0192, Buenos Aires
  - Local Institution - 0193, Mendoza
- Australia (6):
  - Local Institution - 0220, Phillip, Australian Capital Territory
  - Local Institution - 0137, Botany, New South Wales
  - Local Institution - 0133, Westmead, New South Wales
  - Local Institution - 0132, Woolloongabba, Queensland
  - Local Institution - 0211, Hobart, Tasmania
  - Local Institution - 0136, Camberwell, Victoria
- Brazil (7):
  - Local Institution - 0109, Vitória, Espírito Santo
  - Local Institution - 0001, Salvador, Estado de Bahia
  - Local Institution - 0002, Juiz de Fora, Minas Gerais
  - Local Institution - 0219, Curitiba, Paraná
  - Local Institution - 0214, Curitiba, Paraná
  - Local Institution - 0005, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0108, Santo André, São Paulo
- Bulgaria (10):
  - Local Institution - 0255, Plovdiv, Plovdiv
  - Local Institution - 0248, Sofia, Sofia (stolitsa)
  - Local Institution - 0253, Burgas
  - Local Institution - 0249, Plovdiv
  - Local Institution - 0267, Plovdiv
  - Local Institution - 0246, Plovdiv
  - Local Institution - 0247, Plovdiv
  - Local Institution - 0245, Sofia
  - Local Institution - 0259, Sofia
  - Local Institution - 0250, Varna
- Chile (6):
  - Local Institution - 0261, Viña del Mar, Región de Valparaíso
  - Local Institution - 0226, Santiago, Santiago Metropolitan
  - Local Institution - 0099, Santiago, Santiago Metropolitan
  - Local Institution - 0073, Santiago, Santiago Metropolitan
  - Local Institution - 0222, Santiago, Santiago Metropolitan
  - Local Institution - 0111, Santiago, Santiago Metropolitan
- China (8):
  - Local Institution - 0149, Hefei, Anhui
  - Local Institution - 0159, Beijing, Beijing Municipality
  - Local Institution - 0190, Chongqing, Chongqing Municipality
  - Local Institution - 0147, Guangzhou, Guangdong
  - Local Institution - 0143, Shenzhen, Guangdong
  - Local Institution - 0150, Dalian, Liaoning
  - Local Institution - 0146, Shanghai, Shanghai Municipality
  - Local Institution - 0145, Yiwu, Zhejiang
- Colombia (8):
  - Local Institution - 0071, Bucaramanga, Santander Department
  - Local Institution - 0072, Barranquilla
  - Local Institution - 0069, Bogotá
  - Local Institution - 0063, Bogotá
  - Local Institution - 0070, Cali
  - Local Institution - 0094, Medellín
  - Local Institution - 0064, Medellín
  - Local Institution - 0065, Zipaquirá
- Czechia (7):
  - Local Institution - 0225, Prague, Praha 5
  - Local Institution - 0269, Uherské Hradiště, Zlín
  - Local Institution - 0202, Zlín, Zlín
  - Local Institution - 0018, Ostrava
  - Local Institution - 0208, Pardubice
  - Local Institution - 0097, Prague
  - Local Institution - 0017, Prague
- Finland (3):
  - Local Institution - 0089, Kuopio, Northern Savonia
  - Local Institution - 0013, Helsinki
  - Local Institution - 0119, Turku
- France (3):
  - Local Institution - 0077, Chambray-lès-Tours
  - Local Institution - 0075, Montpellier
  - Local Institution - 0074, Paris
- Hungary (8):
  - Local Institution - 0270, Gyula, Bekes County
  - Local Institution - 0049, Székesfehérvár, Fejér
  - Local Institution - 0023, Budapest
  - Local Institution - 0142, Budapest
  - Local Institution - 0026, Budapest
  - Local Institution - 0025, Budapest
  - Local Institution - 0203, Budapest
  - Local Institution - 0068, Zalaegerszeg
- Ireland (4):
  - Local Institution - 0104, Manorhamilton, Leitrim
  - Local Institution - 0101, Dublin
  - Local Institution - 0102, Dublin
  - Local Institution - 0103, Galway
- Italy (4):
  - Local Institution - 0066, Genova
  - Local Institution - 0062, Pavia
  - Local Institution - 0096, Udine
  - Local Institution - 0058, Verona
- Mexico (9):
  - Local Institution - 0056, Saltillo, Coahuila
  - Local Institution - 0254, Guadalajara, Jalisco
  - Local Institution - 0057, Mexico City, Mexico City
  - Local Institution - 0128, San Luis Potosí City, San Luis Potosí
  - Local Institution - 0061, Mérida, Yucatán
  - Local Institution - 0212, Mérida, Yucatán
  - Local Institution - 0060, Chihuahua City
  - Local Institution - 0209, Mexico City
  - Local Institution - 0095, Veracruz
- Poland (27):
  - Local Institution - 0231, Dąbrówka, Greater Poland Voivodeship
  - Local Institution - 0229, Krakow, Lesser Poland Voivodeship
  - Local Institution - 0206, Nowy Targ, Lesser Poland Voivodeship
  - Local Institution - 0244, Wroclaw, Lower Silesian Voivodeship
  - Local Institution - 0232, Lublin, Lublin Voivodeship
  - Local Institution - 0230, Świdnik, Lublin Voivodeship
  - Local Institution - 0233, Nadarzyn, Masovian Voivodeship
  - Local Institution - 0235, Warsaw, Masovian Voivodeship
  - Local Institution - 0243, Warsaw, Masovian Voivodeship
  - Local Institution - 0236, Wołomin, Masovian Voivodeship
  - Local Institution - 0257, Gdansk, Pomeranian Voivodeship
  - Local Institution - 0234, Gdynia, Pomeranian Voivodeship
  - Local Institution - 0241, Częstochowa, Silesian Voivodeship
  - Local Institution - 0252, Katowice, Silesian Voivodeship
  - Local Institution - 0114, Bialystok
  - Local Institution - 0126, Krakow
  - Local Institution - 0127, Krakow
  - Local Institution - 0140, Krakow
  - Local Institution - 0162, Olsztyn
  - Local Institution - 0113, Poznan
  - Local Institution - 0239, Poznan
  - Local Institution - 0112, Poznan
  - Local Institution - 0204, Warsaw
  - Local Institution - 0205, Warsaw
  - Local Institution - 0125, Warsaw
  - Local Institution - 0210, Wroclaw
  - Local Institution - 0238, Lodz, Łódź Voivodeship
- Romania (14):
  - Local Institution - 0090, Bucharest, București
  - Local Institution - 0266, Bucharest, București
  - Local Institution - 0010, Râmnicu Vâlcea, Vâlcea County
  - Local Institution - 0012, Brasov
  - Local Institution - 0167, Bucharest
  - Local Institution - 0260, Bucharest
  - Local Institution - 0263, Bucharest
  - Local Institution - 0184, Bucharest
  - Local Institution - 0011, Cluj-Napoca
  - Local Institution - 0258, Craiova
  - Local Institution - 0262, Iași
  - Local Institution - 0265, Iași
  - Local Institution - 0264, Iași
  - Local Institution - 0091, Timișoara
- Russia (4):
  - Local Institution, Kemerovo
  - Local Institution, Korolyov
  - Local Institution, Saint Petersburg
  - Local Institution, Yaroslavl
- Spain (4):
  - Local Institution - 0021, A Coruña
  - Local Institution - 0022, Córdoba
  - Local Institution - 0019, Madrid
  - Local Institution - 0020, Sabadell
- Taiwan (5):
  - Local Institution - 0123, Kaohsiung City
  - Local Institution - 0121, Tainan
  - Local Institution - 0122, Tainan
  - Local Institution - 0120, Taipei
  - Local Institution - 0124, Taoyuan District
- United Kingdom (3):
  - Local Institution - 0106, Southampton, Hampshire
  - Local Institution - 0116, Harlow
  - Local Institution - 0107, Stoke-on-Trent

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT04908202.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo-Controlled Period - Deucravacitinib 6 mg QD: Participants with Active Psoriatic Arthritis who are naive to biologic disease anti-rheumatic drugs were administered 6 mg of deucravacitinib tablet orally once daily (QD) from Week 1 till Week 16 during Placebo-Controlled treatment period.
- Placebo-Controlled Period - Placebo: Participants with Active Psoriatic Arthritis who are naive to biologic disease anti-rheumatic drugs were administered placebo tablet orally once daily (QD) from Week 1 till Week 16 during Placebo-Controlled treatment period.
- Active Treatment Period - Deucravacitinib 6 mg QD: Participants earlier randomized to Deucravacitinib 6 mg QD arm in Placebo-Controlled period continued to receive 6 mg deucravacitinib tablet orally QD till Week 52 during Active Treatment period.
- Active-Treatment Period - Placebo-Deucravacitinib 6 mg QD: Participants earlier randomized to Placebo arm in Placebo-Controlled period received 6 mg deucravacitinib tablet orally QD till Week 52 during Active Treatment period.
Period: Pre-Treatment Period
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo | Active Treatment Period - Deucravacitinib 6 mg QD | Active-Treatment Period - Placebo-Deucravacitinib 6 mg QD
Started | 336 | 334 | 0 | 0
Completed | 332 | 333 | 0 | 0
Not Completed | 4 | 1 | 0 | 0
Not completed — OTHER REASONS | 3 | 1 | 0 | 0
Not completed — PARTICIPANT WITHDREW CONSENT | 1 | 0 | 0 | 0
Period: Placebo-Controlled Treatment Period
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo | Active Treatment Period - Deucravacitinib 6 mg QD | Active-Treatment Period - Placebo-Deucravacitinib 6 mg QD
Started | 332 | 333 | 0 | 0
Completed | 309 | 306 | 0 | 0
Not Completed | 23 | 27 | 0 | 0
Not completed — Lack of Efficacy | 1 | 2 | 0 | 0
Not completed — Adverse Event | 8 | 6 | 0 | 0
Not completed — PARTICIPANT REQUEST TO DISCONTINUE STUDY TREATMENT | 2 | 3 | 0 | 0
Not completed — PARTICIPANT WITHDREW CONSENT | 4 | 10 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — ADMINISTRATIVE REASONS BY SPONSOR | 0 | 1 | 0 | 0
Not completed — Other reasons | 8 | 4 | 0 | 0
Period: Active Treatment Period
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo | Active Treatment Period - Deucravacitinib 6 mg QD | Active-Treatment Period - Placebo-Deucravacitinib 6 mg QD
Started | 0 | 0 | 309 | 306
Completed | 0 | 0 | 168 | 160
Not Completed | 0 | 0 | 141 | 146
Not completed — OTHER REASONS | 0 | 0 | 1 | 3
Not completed — Lack of Efficacy | 0 | 0 | 4 | 5
Not completed — Adverse Event | 0 | 0 | 5 | 8
Not completed — PARTICIPANT REQUEST TO DISCONTINUE STUDY TREATMENT | 0 | 0 | 2 | 2
Not completed — PARTICIPANT WITHDREW CONSENT | 0 | 0 | 8 | 11
Not completed — Lost to Follow-up | 0 | 0 | 2 | 2
Not completed — POOR/NON-COMPLIANCE | 0 | 0 | 1 | 0
Not completed — ADMINISTRATIVE REASONS BY SPONSOR | 0 | 0 | 1 | 1
Not completed — ONGOING Treatment | 0 | 0 | 117 | 114

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo | Total
Number analyzed (Participants) | 336 | 334 | 670
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (12.52) | 52.3 (12.32) | 52.0 (12.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 164 | 170 | 334
  Male | 172 | 164 | 336
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 101 | 94 | 195
  Not Hispanic or Latino | 165 | 165 | 330
  Unknown or Not Reported | 70 | 75 | 145
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  WHITE | 263 | 279 | 542
  BLACK OR AFRICAN AMERICAN | 4 | 1 | 5
  AMERICAN INDIAN OR ALASKA NATIVE | 17 | 19 | 36
  OTHER | 27 | 21 | 48
  CHINESE | 24 | 14 | 38
  ASIAN OTHER | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With ACR 20 Response at Week 16
Description: The ACR 20 definition of improvement is a 20% improvement over baseline in tender and swollen joint counts (#1 and #2) and a 20% improvement in 3 of the 5 remaining core data set measures (Participant global assessment of pain, participant global assessment of disease activity, physician global assessment of disease activity, participant assessment of physical function, and acute phase reactant value). Baseline value is the last assessment taken prior to first dose of single-blind study medication. The 95% CI is calculated using Clopper-Pearson exact method.
Time Frame: Week 16
Population: Randomized population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 336 | 334
percentage of participants | 54.2 [48.7 to 59.6] | 34.1 [29.1 to 39.5]
Statistical Analysis 1: Comparison: Placebo-Controlled Period - Deucravacitinib 6 mg QD vs Placebo-Controlled Period - Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.29, 95% CI 2-sided [1.67 to 3.13]

2. Secondary Outcome: Change From Baseline in Disease Activity Score 28 C-reactive Protein (DAS28-CRP) at Week 16
Description: DAS28-CRP is a composite of how many joints in the hands (including metacarpophalangeal and proximal interphalangeal joints but excluding DIPs), wrists, elbows, shoulders, and knees are swollen and/or tender out of a total of 28; CRP in the blood to measure the degree of inflammation, and participant global assessment of disease activity. The results are combined to produce the DAS28-CRP score that range from 1.0 to 9.4, which correlates with the extent of disease activity: < 2.6=disease remission; 2.6 - 3.2=low disease activity; 3.2-5.1=moderate disease activity; >5.1=high disease activity. Change from baseline is defined as value at post-baseline visit. A negative change from baseline in DAS28-CRP indicates an improvement.
Time Frame: Baseline and Week 16
Population: Randomized population. Only participants with data available at the timepoint were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 317 | 317
Score on a Scale | -1.4106 (1.13277) | -0.8902 (1.10750)
Statistical Analysis 1: Comparison: Placebo-Controlled Period - Deucravacitinib 6 mg QD vs Placebo-Controlled Period - Placebo; Test type: Superiority; p < 0.0001, ANCOVA; ADJUSTED MEAN DIFFERENCE = -0.5051, 95% CI 2-sided [-0.6709 to -0.3392]

3. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI) at Week 16
Description: HAQ-DI is a patient-reported outcome measure that assesses the degree of difficulty a participant has experienced during the past week in 8 domains of daily living activities: dressing and grooming, arising, eating, walking, hygiene, reach, grip, and other activities. Each activity category consists of 2 to 3 items. For each item in the questionnaire, the level of activity is scored from 0 to 3, with 0 representing "no difficulty," 1 representing "some difficulty," 2 representing "much difficulty," and 3 representing "unable to do." increasing scores for the 8 disability categories indicate increasing level of difficulty. HAQDI is calculated by summing the adjusted categories scores and dividing by the number of categories answered. Change from baseline is defined as value at post-baseline visit. A negative change from baseline in HAQ-DI indicates an improvement.
Time Frame: Baseline and Week 16
Population: Randomized population. Only participants with data available at the timepoint were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 326 | 327
Score on a Scale | -0.4103 (0.52303) | -0.2118 (0.51583)
Statistical Analysis 1: Comparison: Placebo-Controlled Period - Deucravacitinib 6 mg QD vs Placebo-Controlled Period - Placebo; Test type: Superiority; p < 0.0001, ANCOVA; ADJUSTED MEAN DIFFERENCE = -0.1688, 95% CI 2-sided [-0.2442 to -0.0933]

4. Secondary Outcome: Percentage of Participants Meeting Psoriatic Area and Severity Index (PASI) 75 Response at Week 16, in Participants With at Least 3% Body Surface Area (BSA) Involvement and at Least Static Physician's Global Assessment (sPGA) 2 at Baseline
Description: PASI is a measure of the average erythema, induration thickness, and scaling of psoriatic skin lesions (each graded on a 0 to 4 scale), weighted by the area of involvement (head, arms, trunk to groin, and legs to top of buttocks). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. PASI 75 is the number of participants who experience at least a 75% improvement in PASI score as compared with the baseline value. The 95% CI is calculated using Clopper-Pearson exact method.
Time Frame: Week 16
Population: Randomized population with participants with at least 3% body surface area (BSA) Involvement and at least static Physician's Global Assessment (sPGA) 2 at baseline
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 162 | 170
percentage of participants | 51.9 [43.9 to 59.8] | 7.1 [3.7 to 12.0]
Statistical Analysis 1: Comparison: Placebo-Controlled Period - Deucravacitinib 6 mg QD vs Placebo-Controlled Period - Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 14.08, 95% CI 2-sided [7.19 to 27.59]

5. Secondary Outcome: Change From Baseline in the 36-item Short Form (SF-36) Physical Subcomponent Summary (PCS) Score at Week 16
Description: SF-36 is a generic 36-item questionnaire measuring health-related quality of life. The physical subcomponent summary (PCS) consists of these 4 subscales: Physical functioning, Role-physical, Bodily pain, General health. The scores range from 0 to 100, with a higher score indicating better quality of life. The PCS summary scores will be calculated by taking a weighted linear combination of the individual subscales. Change from baseline is defined as value at post-baseline visit. A negative change from baseline in SF-36 PCS indicates an improvement.
Time Frame: Baseline and Week 16
Population: Randomized population. Only participants with data available at the timepoint were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 326 | 327
Score on a Scale | 6.410 (8.2883) | 3.847 (7.2929)
Statistical Analysis 1: Comparison: Placebo-Controlled Period - Deucravacitinib 6 mg QD vs Placebo-Controlled Period - Placebo; Test type: Superiority; p < 0.0001, ANCOVA; ADJUSTED MEAN DIFFERENCE = 6.631, 95% CI 2-sided [3.481 to 9.781]

6. Secondary Outcome: Percentage of Participants Meeting Enthesitis Resolution (Score of 0) Among Participants With Enthesitis at Baseline by Leeds Enthesitis Index (LEI) at Week 16
Description: Percentage of participants meeting enthesitis resolution (score of 0) among participants with enthesitis at Baseline by Leeds Enthesitis Index (LEI). An overall score of 0 to 6 is derived from the presence or absence of tenderness at 6 enthesial sites (right and left: lateral epicondyle, medial femoral condyle, and Achilles tendon insertion) at the time of evaluation. A higher count indicates a greater enthesitis burden.
Time Frame: Week 16
Population: Randomized population with Enthesitis at Baseline by LEI
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 178 | 167
percentage of participants | 48.3 [40.8 to 55.9] | 46.1 [38.4 to 54.0]
Statistical Analysis 1: Comparison: Placebo-Controlled Period - Deucravacitinib 6 mg QD vs Placebo-Controlled Period - Placebo; Test type: Superiority; p = 0.5699, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.74 to 1.75]

7. Secondary Outcome: Percentage of Participants Meeting Achievement of Minimal Disease Activity (MDA) at Week 16
Description: Percentage of participants meeting achievement of MDA where an MDA response is achievement of 5 of 7 following outcomes at Week 16:
  1. Tender joint count <= 1
  2. Swollen joint count <=1
  3. Psoriasis Area and Severity Index (PASI) <= 1 or body surface area (BSA) <= 3%
  4. Patient assessment of psoriatic arthiritis (PsA) pain <= 15
  5. Patient Global Assessment of PsA disease activity <= 20
  6. HAQ-DI <= 0.5
  7. Tender enthesial points <= 1
Time Frame: Week 16
Population: Randomized population. Only participants with available data at the timepoint were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 336 | 334
percentage of participants | 19.0 [15.0 to 23.7] | 10.2 [7.2 to 13.9]
Statistical Analysis 1: Comparison: Placebo-Controlled Period - Deucravacitinib 6 mg QD vs Placebo-Controlled Period - Placebo; Test type: Superiority; p = 0.0012, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.08, 95% CI 2-sided [1.33 to 3.26]

8. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-Fatigue) Score at Week 16
Description: FACIT-Fatigue evaluates a range of self-reported symptoms over the past week, from mild subjective feelings of tiredness to an overwhelming, debilitating, and sustained sense of exhaustion that likely decreases one's ability to execute daily activities and function normally in family or social roles. Fatigue is divided into the experience or symptoms of fatigue (frequency, duration, and intensity) and the impact of fatigue on physical, mental, and social activities. The recall period is 7 days. Each item is rated on a 5-point Likert scale ranging from 0 = "not at all" to 4 = "very much." Sum scores for the 13 items range from 0 through 52, where higher scores indicate less fatigue. Change from baseline is defined as value at post-baseline visit. A negative change from baseline in FACIT-Fatigue indicates an improvement.
Time Frame: Baseline and Week 16
Population: Randomized population. Only participants with data available at the timepoint were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 326 | 326
Score on a Scale | 4.9 (8.84) | 2.2 (8.81)
Statistical Analysis 1: Comparison: Placebo-Controlled Period - Deucravacitinib 6 mg QD vs Placebo-Controlled Period - Placebo; Test type: Superiority; p < 0.0001, ANCOVA; ADJUSTED MEAN DIFFERENCE = 2.6, 95% CI 2-sided [1.4 to 3.9]

9. Secondary Outcome: Percentage of Participants Meeting Dactylitis Resolution at Week 16
Description: Percentage of participants meeting dactylitis resolution at Week 16 among the participants with dactylitis at baseline, where resolution is defined as a tender dactylitis count of 0 in participants with a tender dactylitis count => 1 at baseline. The number of digits in hands and feet with dactylitis will be counted by a blinded assessor.
Time Frame: Week 16
Population: Randomized population. Only participants with tender dactylitis count >=1 at baseline were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 132 | 108
percentage of participants | 59.1 [50.2 to 67.6] | 43.5 [34.0 to 53.4]
Statistical Analysis 1: Comparison: Placebo-Controlled Period - Deucravacitinib 6 mg QD vs Placebo-Controlled Period - Placebo; Test type: Superiority; p = 0.0270, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.80, 95% CI 2-sided [1.07 to 3.03]

10. Secondary Outcome: Change From Baseline in PsA-modified Sharp-van Der Heijde (SvdH) Score at Week 16
Description: The PsA-modified Sharp-van der Heijde (SvdH) score is a radiographic tool used to assess structural joint damage in psoriatic arthritis. It evaluates erosions, joint space narrowing, (sub)luxation, and ankylosis in 52 joints of the hands and feet, including distal interphalangeal joints. Erosions are scored 0-3 and joint space narrowing 0-4. The total score ranges from 0 to 528 (erosions: max 320; joint space narrowing: max 208). Higher scores indicate greater joint damage. Change from baseline reflects progression or improvement; a decrease suggests reduced damage or improvement.
Time Frame: Baseline and Week 16
Population: Randomized population. Only participants with data available at the timepoint were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 245 | 251
Score on a Scale | 0.3980 (2.00852) | 0.5757 (2.73874)
Statistical Analysis 1: Comparison: Placebo-Controlled Period - Deucravacitinib 6 mg QD vs Placebo-Controlled Period - Placebo; Test type: Superiority; p = 0.7194, ANCOVA; ADJUSTED MEAN DIFFERENCE = 0.1596, 95% CI 2-sided [-0.7114 to 1.0306]

11. Secondary Outcome: Percentage of Participants With ACR 20 Response up to Week 16
Description: as for outcome 1
Time Frame: Week 2, 4, 8, 12, and 16
Population: Randomized population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 336 | 334
percentage of participants
  Week 2 | 14.0 [10.5 to 18.2] | 13.8 [10.3 to 17.9]
  Week 4 | 31.5 [26.6 to 36.8] | 19.5 [15.4 to 24.1]
  Week 8 | 42.6 [37.2 to 48.0] | 30.5 [25.6 to 35.8]
  Week 12 | 49.1 [43.6 to 54.6] | 31.1 [26.2 to 36.4]
  Week 16 | 54.2 [48.7 to 59.6] | 34.1 [29.1 to 39.5]

12. Secondary Outcome: Percentage of Participants With ACR 50 Response up to Week 16
Description: The ACR 50 definition of improvement is a 50% improvement over baseline in tender and swollen joint counts (#1 and #2) and a 50% improvement in 3 of the 5 remaining core data set measures (Participant global assessment of pain, participant global assessment of disease activity, physician global assessment of disease activity, participant assessment of physical function, and acute phase reactant value). Baseline value is the last assessment taken prior to first dose of single-blind study medication. The 95% CI is calculated using Clopper-Pearson exact method.
Time Frame: Week 2, 4, 8, 12, and 16
Population: Randomized population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 336 | 334
percentage of participants
  Week 2 | 2.1 [0.8 to 4.2] | 1.2 [0.3 to 3.0]
  Week 4 | 7.7 [5.1 to 11.1] | 3.6 [1.9 to 6.2]
  Week 8 | 17.0 [13.1 to 21.4] | 9.6 [6.6 to 13.3]
  Week 12 | 22.6 [18.3 to 27.5] | 10.8 [7.7 to 14.6]
  Week 16 | 24.7 [20.2 to 29.7] | 13.5 [10.0 to 17.6]

13. Secondary Outcome: Percentage of Participants With ACR 70 Response up to Week 16
Description: The ACR 70 definition of improvement is a 70% improvement over baseline in tender and swollen joint counts (#1 and #2) and a 70% improvement in 3 of the 5 remaining core data set measures (Participant global assessment of pain, participant global assessment of disease activity, physician global assessment of disease activity, participant assessment of physical function, and acute phase reactant value). Baseline value is the last assessment taken prior to first dose of single-blind study medication. The 95% CI is calculated using Clopper-Pearson exact method.
Time Frame: Week 2, 4, 8, 12, and 16
Population: Randomized population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 336 | 334
percentage of participants
  Week 2 | 0.3 [0.0 to 1.6] | 0.0 [0.0 to 1.1]
  Week 4 | 1.8 [0.7 to 3.8] | 0.0 [0.0 to 1.1]
  Week 8 | 5.7 [3.4 to 8.7] | 3.0 [1.4 to 5.4]
  Week 12 | 7.4 [4.9 to 10.8] | 3.6 [1.9 to 6.2]
  Week 16 | 11.6 [8.4 to 15.5] | 5.4 [3.2 to 8.4]

14. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI) up to Week 16
Description: as for outcome 3
Time Frame: Baseline and Week 2, 4, 8, 12, and 16
Population: Randomized population. Only participants with data available at the timepoint were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 327 | 327
Score on a Scale
  Week 2 (n=324, 323): number analyzed (Participants) | 324 | 323
  Week 2 (n=324, 323) | -0.1655 (0.37744) | -0.1250 (0.38243)
  Week 4 (n=325, 326): number analyzed (Participants) | 325 | 326
  Week 4 (n=325, 326) | -0.2412 (0.43862) | -0.1614 (0.39402)
  Week 8 (n=327, 326): number analyzed (Participants) | 327 | 326
  Week 8 (n=327, 326) | -0.3119 (0.50219) | -0.1963 (0.47057)
  Week 12 (n= 326, 327): number analyzed (Participants) | 326 | 327
  Week 12 (n= 326, 327) | -0.3589 (0.49384) | -0.1957 (0.53080)
  Week 16 (n=326, 327): number analyzed (Participants) | 326 | 327
  Week 16 (n=326, 327) | -0.4103 (0.52303) | -0.2118 (0.51583)

15. Secondary Outcome: Percentage of Participants Who Achieve a Clinically Meaningful Improvement in Health Assessment Questionnaire - Disability Index (HAQ-DI) up to Week 16 Among Participants With a HAQ-DI Score ≥0.35 at Baseline
Description: HAQ-DI is a patient-reported outcome measure that assesses the degree of difficulty a participant has experienced during the past week in 8 domains of daily living activities: dressing and grooming, arising, eating, walking, hygiene, reach, grip, and other activities. Each activity category consists of 2 to 3 items. For each item in the questionnaire, the level of activity is scored from 0 to 3, with 0 representing "no difficulty," 1 representing "some difficulty," 2 representing "much difficulty," and 3 representing "unable to do." increasing scores for the 8 disability categories indicate increasing level of difficulty. HAQDI is calculated by summing the adjusted categories scores and dividing by the number of categories answered. Clinically meaningful improvement was defined as ≥0.35improvement from baseline.
Time Frame: Baseline and Week 2, 4, 8, 12, and 16
Population: Randomized population. Only participants with a HAQ-DI score ≥0.35 at Baseline were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 314 | 307
Percentage of Participants
  Week 2 | 28.0 [23.1 to 33.3] | 28.0 [23.1 to 33.4]
  Week 4 | 41.4 [35.9 to 47.1] | 30.9 [25.8 to 36.4]
  Week 8 | 45.5 [39.9 to 51.2] | 34.2 [28.9 to 39.8]
  Week 12 | 49.7 [44.0 to 55.4] | 39.7 [34.2 to 45.5]
  Week 16 | 51.3 [45.6 to 56.9] | 38.8 [33.3 to 44.5]

16. Secondary Outcome: Percentage of Participants Meeting Psoriatic Area and Severity Index (PASI) 75 Response up to Week 16, in Participants With at Least 3% Body Surface Area (BSA) Involvement and at Least Static Physician's Global Assessment (sPGA) 2 at Baseline
Description: as for outcome 4
Time Frame: Week 4, 8, 12 and 16
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 162 | 170
percentage of participants
  Week 4 | 11.7 [7.2 to 17.7] | 6.5 [3.3 to 11.3]
  Week 8 | 31.5 [24.4 to 39.2] | 10.0 [5.9 to 15.5]
  Week 12 | 42.6 [34.9 to 50.6] | 8.8 [5.0 to 14.1]
  Week 16 | 51.9 [43.9 to 59.8] | 7.1 [3.7 to 12.0]

17. Secondary Outcome: Percentage of Participants Meeting Psoriatic Area and Severity Index (PASI) 90 Response up to Week 16, in Participants With at Least 3% Body Surface Area (BSA) Involvement and at Least Static Physician's Global Assessment (sPGA) 2 at Baseline
Description: PASI is a measure of the average erythema, induration thickness, and scaling of psoriatic skin lesions (each graded on a 0 to 4 scale), weighted by the area of involvement (head, arms, trunk to groin, and legs to top of buttocks). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. PASI 90 is the number of participants who experience at least a 90% improvement in PASI score as compared with the baseline value. The 95% CI is calculated using Clopper-Pearson exact method.
Time Frame: Week 4, 8, 12 and 16
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 162 | 170
percentage of participants
  Week 4 | 4.3 [1.8 to 8.7] | 1.8 [0.4 to 5.1]
  Week 8 | 14.8 [9.7 to 21.2] | 1.8 [0.4 to 5.1]
  Week 12 | 20.4 [14.5 to 27.4] | 3.5 [1.3 to 7.5]
  Week 16 | 25.3 [18.8 to 32.7] | 1.8 [0.4 to 5.1]

18. Secondary Outcome: Percentage of Participants Meeting Psoriatic Area and Severity Index (PASI) 100 Response up to Week 16, in Participants With at Least 3% Body Surface Area (BSA) Involvement and at Least Static Physician's Global Assessment (sPGA) 2 at Baseline
Description: PASI is a measure of the average erythema, induration thickness, and scaling of psoriatic skin lesions (each graded on a 0 to 4 scale), weighted by the area of involvement (head, arms, trunk to groin, and legs to top of buttocks). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. PASI 100 is the number of participants who experience at least a 100% improvement in PASI score as compared with the baseline value. The 95% CI is calculated using Clopper-Pearson exact method.
Time Frame: Week 4, 8, 12 and 16
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 162 | 170
percentage of participants
  Week 4 | 1.9 [0.4 to 5.3] | 1.2 [0.1 to 4.2]
  Week 8 | 8.0 [4.3 to 13.3] | 0.6 [0.0 to 3.2]
  Week 12 | 11.1 [6.7 to 17.0] | 1.8 [0.4 to 5.1]
  Week 16 | 14.2 [9.2 to 20.5] | 1.8 [0.4 to 5.1]

19. Secondary Outcome: Change From Baseline in the 36-item Short Form (SF-36) Physical Subcomponent Summary (PCS) Score up to Week 16
Description: SF-36 is a generic 36-item questionnaire measuring health-related quality of life. The physical subcomponent summary (PCS) consists of these 4 subscales: Physical functioning, Role-physical, Bodily pain, General health. The scores range from 0 to 100, with a higher score indicating poor quality of life. The PCS summary scores will be calculated by taking a weighted linear combination of the individual subscales. Change from baseline is defined as value at post-baseline visit. A negative change from baseline in SF-36 PCS indicates an improvement.
Time Frame: Baseline and Week 4, 12 and 16
Population: Randomized population. Only participants with data available at the timepoint were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 326 | 327
Score on a Scale
  Week 4: number analyzed (Participants) | 325 | 325
  Week 4 | 3.760 (6.2768) | 3.326 (5.7315)
  Week 12: number analyzed (Participants) | 325 | 325
  Week 12 | 6.021 (7.5809) | 3.916 (7.6614)
  Week 16 | 6.410 (8.2883) | 3.847 (7.2929)

20. Secondary Outcome: Percentage of Participants Meeting Enthesitis Resolution (Score of 0) Among Participants With Enthesitis at Baseline by Leeds Enthesitis Index (LEI) up to Week 16
Description: as for outcome 6
Time Frame: Week 4, 8, 12 and 16
Population: Randomized population with Enthesitis at Baseline by LEI
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 178 | 167
percentage of participants
  Week 4 | 31.5 [24.7 to 38.8] | 32.9 [25.9 to 40.6]
  Week 8 | 44.4 [37.0 to 52.0] | 47.9 [40.1 to 55.8]
  Week 12 | 47.2 [39.7 to 54.8] | 50.3 [42.5 to 58.1]
  Week 16 | 48.3 [40.8 to 55.9] | 46.1 [38.4 to 54.0]

21. Secondary Outcome: Percentage of Participants Meeting Enthesitis Resolution (Score of 0) Among Participants With Enthesitis at Baseline by Spondyloarthritis Research Consortium of Canada (SPARCC) up to Week 16
Description: Percentage of participants meeting enthesitis resolution (score of 0) among participants with enthesitis at Baseline by SPARCC. The SPARCC Enthesitis Index has a 0 to 16 score that is derived from the evaluation of 8 locations: the greater trochanter (right [R]/left [L]), quadriceps tendon insertion into the patella (R/L), patellar ligament insertion into the patella and tibial tuberosity (R/L), Achilles tendon insertion (R/L), plantar fascia insertion (R/L), medial and lateral epicondyles (R/L), and supraspinatus insertion (R/L). A higher count indicates a higher enthesitis burden based on the current evaluation.
Time Frame: Week 4, 8, 12 and 16
Population: Randomized population with Enthesitis at Baseline by SPARCC
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 216 | 211
percentage of participants
  Week 4 | 19.4 [14.4 to 25.4] | 25.6 [19.8 to 32.0]
  Week 8 | 34.7 [28.4 to 41.5] | 30.8 [24.6 to 37.5]
  Week 12 | 36.6 [30.1 to 43.4] | 34.6 [28.2 to 41.4]
  Week 16 | 45.8 [39.1 to 52.7] | 34.1 [27.8 to 40.9]

22. Secondary Outcome: Percentage of Participants Meeting Achievement of Minimal Disease Activity (MDA) up to Week 16
Description: as for outcome 7
Time Frame: Week 4, 8, 12, and 16
Population: Randomized population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 336 | 334
percentage of participants
  Week 4 | 6.0 [3.7 to 9.0] | 3.0 [1.4 to 5.4]
  Week 8 | 10.1 [7.1 to 13.9] | 6.6 [4.2 to 9.8]
  Week 12 | 14.0 [10.5 to 18.2] | 7.2 [4.7 to 10.5]
  Week 16 | 19.0 [15.0 to 23.7] | 10.2 [7.2 to 13.9]

23. Secondary Outcome: Change From Baseline in the 36-item Short Form (SF-36) Mental Component Summary (MCS) Score up to Week 16
Description: SF-36 is a generic 36-item questionnaire measuring health-related quality of life. The mental component summary (MCS) of the SF-36 consists of these 4 subscales: Vitality, Social functioning, Role-emotional, Mental health. The scores range from 0 to 100, with a higher score indicating poor quality of life. The MCS summary scores will be calculated by taking a weighted linear combination of the individual subscales. Change from baseline is defined as value at post-baseline visit. A negative change from baseline in SF-36 MCS indicates an improvement.
Time Frame: Baseline and Week 4, 12 and 16
Population: Randomized population. Only participants with data available at the timepoint were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 326 | 327
Score on a Scale
  Week 4: number analyzed (Participants) | 325 | 325
  Week 4 | 0.814 (7.5082) | 0.634 (7.3796)
  Week 12: number analyzed (Participants) | 325 | 325
  Week 12 | 2.056 (8.4206) | 0.034 (8.3926)
  Week 16 | 2.588 (8.3442) | 0.358 (8.1559)

24. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-Fatigue) Score up to Week 16
Description: as for outcome 8
Time Frame: Baseline and Week 2, 4, 8, 12 and 16
Population: Randomized population. Only participants with data available at the timepoint were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 327 | 327
Score on a Scale
  Week 2: number analyzed (Participants) | 324 | 323
  Week 2 | 2.2 (7.31) | 2.3 (6.52)
  Week 4: number analyzed (Participants) | 325 | 325
  Week 4 | 2.5 (7.48) | 2.3 (7.67)
  Week 8: number analyzed (Participants) | 327 | 326
  Week 8 | 4.5 (8.68) | 2.8 (9.64)
  Week 12: number analyzed (Participants) | 326 | 327
  Week 12 | 4.3 (8.98) | 1.8 (8.97)
  Week 16: number analyzed (Participants) | 326 | 326
  Week 16 | 4.9 (8.84) | 2.2 (8.81)

25. Secondary Outcome: Percentage of Participants Meeting Dactylitis Resolution up to Week 16
Description: as for outcome 9
Time Frame: Week 4, 8, 12 and 16
Population: Randomized population. Only participants with tender dactylitis count >=1 at baseline were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 132 | 108
percentage of participants
  Week 4 | 36.4 [28.2 to 45.2] | 33.3 [24.6 to 43.1]
  Week 8 | 44.7 [36.0 to 53.6] | 43.5 [34.0 to 53.4]
  Week 12 | 54.5 [45.7 to 63.2] | 48.1 [38.4 to 58.0]
  Week 16 | 59.1 [50.2 to 67.6] | 43.5 [34.0 to 53.4]

26. Secondary Outcome: Change From Baseline in Psoriatic Arthritis Impact of Disease (PsAID) 12 Score up to Week 16
Description: The Psoriatic Arthritis Impact of Disease (PsAID) is a 12-item self-report that measures PsA symptoms and impact of disease. Each item is scored on a 0 to 10 numeric rating scale with a 1-week recall period. The PsAID has a total score, with a higher value indicating worse health. Change from baseline is defined as value at post-baseline visit. A negative change from baseline in PsAID indicates an improvement.
Time Frame: Baseline and Week 2, 4, 8, 12 and 16
Population: Randomized population. Only participants with data available at the timepoint were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 327 | 327
Score on a Scale
  Week 2: number analyzed (Participants) | 324 | 323
  Week 2 | -0.807 (1.3327) | -0.652 (1.2524)
  Week 4: number analyzed (Participants) | 325 | 325
  Week 4 | -1.164 (1.5433) | -0.836 (1.5580)
  Week 8: number analyzed (Participants) | 327 | 326
  Week 8 | -1.545 (1.9037) | -0.991 (1.9281)
  Week 12: number analyzed (Participants) | 326 | 327
  Week 12 | -1.761 (2.0074) | -0.883 (1.9677)
  Week 16: number analyzed (Participants) | 326 | 327
  Week 16 | -1.851 (2.0440) | -1.015 (1.9955)

27. Secondary Outcome: Change From Baseline in Disease Activity Index for Psoriatic Arthritis (DAPSA) Score up to Week 16
Description: The Disease Activity Index for Psoriatic Arthritis Score is a composite measure to assess peripheral joint involvement that is based upon numerical summation of 5 variables of disease activity: tender joint count (0-68), swollen joint count (0-66), Participant Global Assessment of Disease Activity (0 to 10 cm VAS, 0= excellent and 10= poor), Participant Global Assessment of Pain (0 to 10 centimeter [cm] visual analog scale (VAS), 0= no pain, 10= worst possible pain), and C-reactive protein. The DAPSA score ranges from 0 to 154, with a higher score indicating more disease activity. Change from baseline is defined as value at post-baseline visit. A negative change from baseline in DAPSA indicates an improvement.
Time Frame: Baseline and Week 2, 4, 8, 12 and 16
Population: Randomized population. Only participants with data available at the timepoint were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 325 | 323
Score on a Scale
  Week 2: number analyzed (Participants) | 322 | 318
  Week 2 | -7.6211 (13.23221) | -7.0045 (11.71166)
  Week 4: number analyzed (Participants) | 324 | 321
  Week 4 | -12.5643 (14.38734) | -10.1201 (13.64766)
  Week 8 | -16.6770 (16.71038) | -12.3610 (15.70632)
  Week 12: number analyzed (Participants) | 323 | 321
  Week 12 | -19.8346 (17.22613) | -13.2671 (17.41524)
  Week 16: number analyzed (Participants) | 317 | 317
  Week 16 | -20.7263 (18.08249) | -13.4075 (17.31116)

28. Secondary Outcome: Percentage of Participants With Achievement of Disease Activity Index for Psoriatic Arthritis (DAPSA) Low Disease Activity Response up to Week 16
Description: The Disease Activity Index for Psoriatic Arthritis Score is a composite measure to assess peripheral joint involvement that is based upon numerical summation of 5 variables of disease activity: tender joint count (0-68), swollen joint count (0-66), Participant Global Assessment of Disease Activity (0 to 10 cm VAS, 0= excellent and 10= poor), Participant Global Assessment of Pain (0 to 10 centimeter [cm] visual analog scale (VAS), 0= no pain, 10= worst possible pain), and C-reactive protein. A higher DAPSA score indicated more active disease activity.
Time Frame: Baseline and Week 2, 4, 8, 12 and 16
Population: Randomized population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 336 | 334
percentage of participants
  Week 2 | 6.5 [4.1 to 9.7] | 4.5 [2.5 to 7.3]
  Week 4 | 13.7 [10.2 to 17.8] | 9.9 [6.9 to 13.6]
  Week 8 | 21.4 [17.2 to 26.2] | 16.5 [12.7 to 20.9]
  Week 12 | 28.9 [24.1 to 34.0] | 17.4 [13.5 to 21.9]
  Week 16 | 26.2 [21.6 to 31.2] | 18.9 [14.8 to 23.5]

29. Secondary Outcome: Percentage of Participants With Achievement of Disease Activity Index for Psoriatic Arthritis (DAPSA) Disease Remission up to Week 16
Description: The Disease Activity Index for Psoriatic Arthritis Score is a composite measure to assess peripheral joint involvement that is based upon numerical summation of 5 variables of disease activity: tender joint count (0-68), swollen joint count (0-66), Participant Global Assessment of Disease Activity (0 to 10 cm VAS, 0= excellent and 10= poor), Participant Global Assessment of Pain (0 to 10 centimeter [cm] visual analog scale (VAS), 0= no pain, 10= worst possible pain), and C-reactive protein. A higher DAPSA score indicated more active disease activity. A score 0 signifies remission.
Time Frame: Baseline and Week 2, 4, 8, 12 and 16
Population: Randomized population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 336 | 334
percentage of participants
  Week 2 | 0.3 [0.0 to 1.6] | 0.0 [0.0 to 1.1]
  Week 4 | 1.5 [0.5 to 3.4] | 0.6 [0.1 to 2.1]
  Week 8 | 3.0 [1.4 to 5.4] | 1.8 [0.7 to 3.9]
  Week 12 | 5.7 [3.4 to 8.7] | 1.8 [0.7 to 3.9]
  Week 16 | 8.6 [5.9 to 12.2] | 2.7 [1.2 to 5.1]

30. Secondary Outcome: Percentage of Participants Meeting Achievement of Physician Global Assessment-Fingernails (PGA-F) of 0/1 up to Week 16
Description: The PGA-F is a 5-point scale used to assess fingernails separately for nail bed signs and nail matrix signs of disease. A global score of between 0 indicating clear, and 4 indicating severe. The overall condition of the fingernails is rated on a 5-point scale: 0 = clear, 1 = minimal, 2 = mild, 3 = moderate, and 4 = severe.
Time Frame: Week 2, 4, 8, 12 and 16
Population: Randomized population. Only participants with a baseline PGA-F score of ≥3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 71 | 61
percentage of participants
  Week 4 | 12.7 [6.0 to 22.7] | 6.6 [1.8 to 15.9]
  Week 8 | 19.7 [11.2 to 30.9] | 16.4 [8.2 to 28.1]
  Week 12 | 16.9 [9.0 to 27.7] | 21.3 [11.9 to 33.7]
  Week 16 | 23.9 [14.6 to 35.5] | 14.8 [7.0 to 26.2]

31. Secondary Outcome: Change From Baseline in Disease Activity Score 28 C-reactive Protein (DAS28-CRP) up to Week 16
Description: as for outcome 2
Time Frame: Baseline and Week 2, 4, 8, 12 and 16
Population: Randomized population. Only participants with data available at the timepoint were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 325 | 323
Score on a Scale
  Week 2: number analyzed (Participants) | 322 | 318
  Week 2 | -0.4028 (0.77126) | -0.4006 (0.70508)
  Week 4: number analyzed (Participants) | 324 | 321
  Week 4 | -0.7655 (0.90092) | -0.6468 (0.82146)
  Week 8 | -1.0820 (1.02041) | -0.7727 (0.99752)
  Week 12: number analyzed (Participants) | 323 | 321
  Week 12 | -1.3360 (1.13745) | -0.8450 (1.09776)
  Week 16: number analyzed (Participants) | 317 | 317
  Week 16 | -1.4106 (1.13277) | -0.8902 (1.10750)

32. Secondary Outcome: Percentage of Participants Meeting Disease Activity Score 28 C-reactive Protein (DAS28-CRP) Low Disease Activity Response up to Week 16
Description: DAS28-CRP is a composite of how many joints in the hands (including metacarpophalangeal and proximal interphalangeal joints but excluding DIPs), wrists, elbows, shoulders, and knees are swollen and/or tender out of a total of 28; CRP in the blood to measure the degree of inflammation, and participant global assessment of disease activity. The results are combined to produce the DAS28-CRP score that range from 1.0 to 9.4, which correlates with the extent of disease activity: < 2.6=disease remission; 2.6 - 3.2=low disease activity; 3.2-5.1=moderate disease activity; >5.1=high disease activity.
Time Frame: Week 2, 4, 8, 12 and 16
Population: Randomized population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 336 | 334
percentage of participants
  Week 2 | 5.4 [3.2 to 8.3] | 4.8 [2.8 to 7.7]
  Week 4 | 9.8 [6.9 to 13.5] | 6.0 [3.7 to 9.1]
  Week 8 | 11.3 [8.1 to 15.2] | 9.3 [6.4 to 12.9]
  Week 12 | 14.3 [10.7 to 18.5] | 11.7 [8.4 to 15.6]
  Week 16 | 15.2 [11.5 to 19.5] | 8.1 [5.4 to 11.5]

33. Secondary Outcome: Percentage of Participants Meeting Disease Activity Score 28 C-reactive Protein (DAS28-CRP) Disease Remission up to Week 16
Description: as for outcome 32
Time Frame: Week 2, 4, 8, 12 and 16
Population: Randomized population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 336 | 334
percentage of participants
  Week 2 | 2.1 [0.8 to 4.2] | 2.1 [0.8 to 4.3]
  Week 4 | 8.0 [5.4 to 11.5] | 5.4 [3.2 to 8.4]
  Week 8 | 14.9 [11.3 to 19.1] | 8.7 [5.9 to 12.2]
  Week 12 | 20.8 [16.6 to 25.6] | 9.0 [6.1 to 12.6]
  Week 16 | 22.3 [18.0 to 27.2] | 13.8 [10.3 to 17.9]

34. Secondary Outcome: Change From Baseline in Psoriatic Arthritis Disease Activity Score (PASDAS) up to Week 16
Description: The Psoriatic Arthritis Disease Activity Score (PASDAS) is a composite measure calculated from the Physician Global Assessment of PsA, the Participant Global Assessment of Disease Activity, the Short Form-36 PCS, the swollen joint count, the tender joint count, the Enthesitis (LEI), the Dactylitis (LDI) (Basic), and the High-sensitivity C-reactive protein (hsCRP). The range of PASDAS is 0-10. Higher score means more active disease. Change from baseline is defined as value at post-baseline visit. A negative change from baseline indicates an improvement.
Time Frame: Baseline and Week 4, 12 and 16
Population: Randomized population. Only participants with data available at the timepoint were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 317 | 316
Score on a Scale
  Week 4 | -1.0405 (1.03004) | -0.8258 (0.97038)
  Week 12: number analyzed (Participants) | 314 | 315
  Week 12 | -1.7675 (1.37563) | -1.0780 (1.33036)
  Week 16: number analyzed (Participants) | 313 | 314
  Week 16 | -1.9064 (1.45258) | -1.1026 (1.31166)

35. Secondary Outcome: Change From Baseline in Modified Composite Psoriatic Disease Activity Index (mCPDAI) up to Week 16
Description: Four domains are used to calculate the modified Composite Psoriatic Disease Activity Index (mCPDAI): joints (66 swollen joint count and 68 tender joint count; Health Assessment Questionnaire), skin (PASI and DLQI), dactylitis (a simple count of each digit involved), and enthesitis (number of tendons/fascia insertion sites showing enthesitis scored from 0 to 4, based on palpation of Achilles tendon and bilateral plantar fasciae insertion). The mCPDAI is scored using a 4 point scale from 0 (no disease activity) to 3 (most severe disease activity), giving an mCPDAI score range of 0 through 12. A higher score indicates more active disease activity. Change from baseline is defined as value at post-baseline visit. A negative change from baseline indicates an improvement.
Time Frame: Baseline and Week 4, 8, 12 and 16
Population: Randomized population. Only participants with data available at the timepoint were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 325 | 326
Score on a Scale
  Week 4: number analyzed (Participants) | 323 | 322
  Week 4 | -1.2 (1.81) | -0.8 (1.61)
  Week 8: number analyzed (Participants) | 325 | 323
  Week 8 | -1.7 (2.09) | -1.2 (1.89)
  Week 12: number analyzed (Participants) | 324 | 323
  Week 12 | -2.1 (2.16) | -1.3 (2.01)
  Week 16: number analyzed (Participants) | 323 | 326
  Week 16 | -2.2 (2.22) | -1.3 (1.96)

36. Secondary Outcome: Percentage of Participants With Achievement of Psoriatic Arthritis Response Criteria (PsARC) up to Week 16
Description: The Psoriatic Arthritis Response Criteria (PsARC) consists of 4 measurements: tender joint count, swollen joint count, Physician Global Assessment of PsA, and Participant Global Assessment of Disease Activity. In order to be classified as a PsARC responder, participants must achieve improvement in 2 of 4 measures, 1 of which must be joint pain or swelling, without worsening in any measure. Improvement in each of the measures is defined below: 1) Decrease of ≥ 30% in tender joint counts; 2) Decrease of ≥ 30% in swollen joint counts; 3) Decrease of ≥ 20% in Physician Global Assessment of PsA; 4) Decrease of ≥ 20% in Participant's Global Assessment of Disease Activity
Time Frame: Week 2, 4, 8, 12 and 16
Population: Randomized population. Only participants with data available at the timepoint were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 336 | 334
percentage of participants
  Week 2 | 25.9 [21.3 to 30.9] | 21.9 [17.5 to 26.7]
  Week 4 | 47.0 [41.6 to 52.5] | 31.1 [26.2 to 36.4]
  Week 8 | 51.5 [46.0 to 56.9] | 41.3 [36.0 to 46.8]
  Week 12 | 55.4 [49.9 to 60.8] | 39.8 [34.5 to 45.3]
  Week 16 | 62.5 [57.1 to 67.7] | 40.1 [34.8 to 45.6]

37. Secondary Outcome: Percentage of Participants Meeting Achievement of Improvement of Bath Ankylosing Spondylitis Disease Activity (BASDAI) Score up to Week 16
Description: BASDAI consists of a 0 to 10 scale measuring discomfort, pain, and fatigue in response to 6 questions pertaining to the 5 major symptoms of ankylosing spondylitis: 1) Fatigue (medical); 2) Spinal pain; 3) Joint pain and swelling; 4) Areas of localized tenderness; 5) Morning stiffness duration; 6) Morning stiffness severity. A higher count indicates worse disease. Each individual question response is scaled to a 0-10 score by dividing by 10, and the BASDAI is derived using the following formula: BASDAI = ((Q1 + Q2 + Q3 + Q4) + ((Q5 + Q6) / 2)) / 5
Time Frame: Week 2, 4, 8, 12 and 16
Population: Randomized population. Only participants with data available at the timepoint were analyzed. with spondylitis in addition to peripheral joint involvement as their presentation of PsA were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 55 | 49
percentage of participants
  Week 2 | 7.3 [2.0 to 17.6] | 6.1 [1.3 to 16.9]
  Week 4 | 10.9 [4.1 to 22.2] | 16.3 [7.3 to 29.7]
  Week 8 | 18.2 [9.1 to 30.9] | 14.3 [5.9 to 27.2]
  Week 12 | 25.5 [14.7 to 39.0] | 16.3 [7.3 to 29.7]
  Week 16 | 25.5 [14.7 to 39.0] | 14.3 [5.9 to 27.2]

38. Secondary Outcome: Percentage of Participants Meeting Achievement of Total PsA-modified SvdH Scores Response of <= 0 at Week 16
Description: The PsA-modified Sharp-van der Heijde (SvdH) score is a radiographic tool used to assess structural joint damage in psoriatic arthritis. It evaluates erosions, joint space narrowing, (sub)luxation, and ankylosis in 52 joints of the hands and feet, including distal interphalangeal joints. Erosions are scored 0-3 and joint space narrowing 0-4. The total score ranges from 0 to 528 (erosions: max 320; joint space narrowing: max 208). Higher scores indicate greater joint damage.
Time Frame: Week 16
Population: Randomized population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 336 | 334
percentage of participants | 59.5 [54.1 to 64.8] | 53.9 [48.4 to 59.3]

39. Secondary Outcome: Percentage of Participants Meeting Achievement of Total PsA-modified SvdH Scores Response of <= 0.5 at Week 16
Description: as for outcome 38
Time Frame: Week 16
Population: Randomized population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 336 | 334
percentage of participants | 62.8 [57.4 to 68.0] | 60.5 [55.0 to 65.8]

40. Secondary Outcome: Percentage of Participants Meeting Achievement of Total PsA-modified SvdH Scores Response of <= Smallest Detectable Change (SDC) at Week 16
Description: The PsA-modified Sharp-van der Heijde (SvdH) score is a radiographic tool used to assess structural joint damage in psoriatic arthritis. It evaluates erosions, joint space narrowing, (sub)luxation, and ankylosis in 52 joints of the hands and feet, including distal interphalangeal joints. Erosions are scored 0-3 and joint space narrowing 0-4. The total score ranges from 0 to 528 (erosions: max 320; joint space narrowing: max 208). Higher scores indicate greater joint damage. SDC is calculated as 1.96* standard deviation of the paired differences of change from baseline/ square root of (2*k); k is the number of reviewers and is default to 2 in this study.
Time Frame: Week 16
Population: Randomized population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 336 | 334
percentage of participants | 67.6 [62.3 to 72.5] | 66.2 [60.8 to 71.2]

41. Secondary Outcome: Percentage of Participants Meeting Achievement of Total PsA-modified SvdH Erosion Scores Response of <= 0 at Week 16
Description: as for outcome 38
Time Frame: Week 16
Population: Randomized population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 336 | 334
percentage of participants | 60.4 [55.0 to 65.7] | 56.6 [51.1 to 62.0]

42. Secondary Outcome: Percentage of Participants Meeting Achievement of Total PsA-modified SvdH Erosion Scores Response of <= 0.5 at Week 16
Description: as for outcome 38
Time Frame: Week 16
Population: Randomized population. Only participants with data available at the timepoint were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 336 | 334
percentage of participants | 64.3 [58.9 to 69.4] | 62.9 [57.4 to 68.1]

43. Secondary Outcome: Percentage of Participants Meeting Achievement of Total PsA-modified SvdH Erosion Scores Response of <= SDC at Week 16
Description: as for outcome 40
Time Frame: Week 16
Population: Randomized population. Only participants with data available at the timepoint were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 336 | 334
percentage of participants | 66.7 [61.3 to 71.7] | 66.8 [61.4 to 71.8]

44. Secondary Outcome: Percentage of Participants Meeting Achievement of Total PsA-modified SvdH Joint Space Narrowing (JSN) Scores Response of <= 0 at Week 16
Description: as for outcome 38
Time Frame: Week 16
Population: Randomized population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 336 | 334
percentage of participants | 67.6 [62.3 to 72.5] | 64.4 [59.0 to 69.5]

45. Secondary Outcome: Percentage of Participants Meeting Achievement of Total PsA-modified SvdH Joint Space Narrowing (JSN) Scores Response of <= 0.5 at Week 16
Description: as for outcome 38
Time Frame: Week 16
Population: Randomized population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 336 | 334
percentage of participants | 70.5 [65.3 to 75.4] | 68.9 [63.6 to 73.8]

46. Secondary Outcome: Percentage of Participants Meeting Achievement of Total PsA-modified SvdH Joint Space Narrowing (JSN) Scores Response of <= SDC at Week 16
Description: as for outcome 40
Time Frame: Week 16
Population: Randomized population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 336 | 334
percentage of participants | 70.5 [65.3 to 75.4] | 68.9 [63.6 to 73.8]

47. Secondary Outcome: Change From Baseline in PsA-modified SvdH Erosion Scores Response at Week 16
Description: as for outcome 38
Time Frame: Baseline and Week 16
Population: Randomized population. Only participants with data available at the timepoint were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 245 | 251
Score on a Scale | 0.32 (1.417) | 0.37 (1.326)

48. Secondary Outcome: Change From Baseline in PsA-modified SvdH JSN Scores Response at Week 16
Description: as for outcome 38
Time Frame: Baseline and Week 16
Population: Randomized population. Only participants with data available at the timepoint were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 245 | 251
Score on a Scale | 0.09 (0.703) | 0.14 (0.485)

49. Secondary Outcome: Change From Baseline in the 36-item Short Form (SF-36) Physical Subcomponent Summary Score up to Week 16
Description: SF-36 is a generic 36-item questionnaire measuring health-related quality of life. The physical sub component is one of the 4 subscales of PCS. The physical subcomponent scores will be calculated by taking a weighted linear combination of the individual question. The score ranges from 0 to 100, with higher values indication poor quality of life. Change from baseline is defined as value at post-baseline visit. A negative change from baseline in SF-36 physical sub-component indicates an improvement.
Time Frame: Baseline and Week 4, 12 and 16
Population: Randomized population. Only participants with data available at the timepoint were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 326 | 327
Score on a Scale
  Week 4: number analyzed (Participants) | 325 | 325
  Week 4 | 7.923 (17.9483) | 6.908 (17.0306)
  Week 12: number analyzed (Participants) | 325 | 325
  Week 12 | 13.615 (20.5725) | 7.784 (22.4709)
  Week 16 | 15.414 (22.3930) | 8.226 (22.1449)

50. Secondary Outcome: Change From Baseline in the 36-item Short Form (SF-36) Role Activity Subcomponent Summary Score up to Week 16
Description: SF-36 is a generic 36-item questionnaire measuring health-related quality of life. The role activity sub component is one of the 4 subscales of PCS. The role activity subcomponent scores will be calculated by taking a weighted linear combination of the individual question. The score ranges from 0 to 100, with higher values indication poor quality of life. Change from baseline is defined as value at post-baseline visit. A negative change from baseline in SF-36 role activity indicates an improvement.
Time Frame: Baseline and Week 4, 12 and 16
Population: Randomized population. Only participants with data available at the timepoint were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 326 | 327
Score on a Scale
  Week 4: number analyzed (Participants) | 325 | 325
  Week 4 | 6.962 (20.6963) | 7.058 (18.7454)
  Week 12: number analyzed (Participants) | 325 | 325
  Week 12 | 13.096 (22.7372) | 8.365 (21.1286)
  Week 16 | 13.152 (23.6370) | 7.913 (20.8035)

51. Secondary Outcome: Change From Baseline in the 36-item Short Form (SF-36) Bodily Pain Subcomponent Summary Score up to Week 16
Description: SF-36 is a generic 36-item questionnaire measuring health-related quality of life. The bodily pain sub component is one of the 4 subscales of PCS. The bodily pain subcomponent scores will be calculated by taking a weighted linear combination of the individual question. The score ranges from 0 to 100, with higher values indication poor quality of life. Change from baseline is defined as value at post-baseline visit. A negative change from baseline in SF-36 bodily pain subcomponent indicates an improvement.
Time Frame: Baseline and Week 4, 12 and 16
Population: Randomized population. Only participants with data available at the timepoint were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 326 | 327
Score on a Scale
  Week 4: number analyzed (Participants) | 325 | 325
  Week 4 | 10.0 (16.52) | 8.5 (15.47)
  Week 12: number analyzed (Participants) | 325 | 325
  Week 12 | 16.6 (20.96) | 9.4 (19.66)
  Week 16 | 18.2 (21.83) | 10.0 (18.85)

52. Secondary Outcome: Change From Baseline in the 36-item Short Form (SF-36) General Health Perceptions Subcomponent Summary Score up to Week 16
Description: SF-36 is a generic 36-item questionnaire measuring health-related quality of life. The general health perceptions sub component is one of the 4 subscales of PCS. The general health perceptions subcomponent scores will be calculated by taking a weighted linear combination of the individual question. The score ranges from 0 to 100, with higher values indication poor quality of life. Change from baseline is defined as value at post-baseline visit. A negative change from baseline in SF-36 general health perceptions subcomponent indicates an improvement.
Time Frame: Baseline and Week 4, 12 and 16
Population: Randomized population. Only participants with data available at the timepoint were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 326 | 327
Score on a Scale
  Week 4: number analyzed (Participants) | 325 | 325
  Week 4 | 6.1 (12.95) | 5.1 (13.35)
  Week 12: number analyzed (Participants) | 325 | 325
  Week 12 | 8.4 (15.13) | 4.8 (15.02)
  Week 16 | 8.9 (16.00) | 4.6 (14.85)

53. Secondary Outcome: Change From Baseline in the 36-item Short Form (SF-36) Vitality Subcomponent Score up to Week 16
Description: SF-36 is a generic 36-item questionnaire measuring health-related quality of life. The vitality subcomponent is one of the 4 subscales of MCS. The vitality subcomponent scores will be calculated by taking a weighted linear combination of the individual question. The score ranges from 0 to 100, with higher values indication poor quality of life. Change from baseline is defined as value at post-baseline visit. A negative change from baseline in SF-36 vitality subcomponent indicates an improvement.
Time Frame: Baseline and Week 4, 12 and 16
Population: Randomized population. Only participants with data available at the timepoint were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 326 | 327
Score on a Scale
  Week 4: number analyzed (Participants) | 325 | 325
  Week 4 | 4.558 (14.6829) | 4.327 (14.3971)
  Week 12: number analyzed (Participants) | 325 | 325
  Week 12 | 8.442 (17.9283) | 4.308 (17.6763)
  Week 16 | 9.682 (16.4474) | 4.893 (17.5265)

54. Secondary Outcome: Change From Baseline in the 36-item Short Form (SF-36) Social Subcomponent Score up to Week 16
Description: SF-36 is a generic 36-item questionnaire measuring health-related quality of life. The social subcomponent is one of the 4 subscales of MCS. The social subcomponent scores will be calculated by taking a weighted linear combination of the individual question. The score ranges from 0 to 100, with higher values indication poor quality of life. Change from baseline is defined as value at post-baseline visit. A negative change from baseline in SF-36 social subcomponent indicates an improvement.
Time Frame: Baseline and Week 4, 12 and 16
Population: Randomized population. Only participants with data available at the timepoint were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 326 | 327
Score on a Scale
  Week 4: number analyzed (Participants) | 325 | 325
  Week 4 | 6.69 (20.610) | 4.62 (20.737)
  Week 12: number analyzed (Participants) | 325 | 325
  Week 12 | 11.96 (23.990) | 4.88 (22.539)
  Week 16 | 13.80 (22.960) | 4.74 (23.303)

55. Secondary Outcome: Change From Baseline in the 36-item Short Form (SF-36) Mental Health Subcomponent Score up to Week 16
Description: SF-36 is a generic 36-item questionnaire measuring health-related quality of life. The mental health subcomponent is one of the 4 subscales of MCS. The mental health subcomponent scores will be calculated by taking a weighted linear combination of the individual question. The score ranges from 0 to 100, with higher values indication poor quality of life. Change from baseline is defined as value at post-baseline visit. A negative change from baseline in SF-36 mental health subcomponent indicates an improvement.
Time Frame: Baseline and Week 4, 12 and 16
Population: Randomized population. Only participants with data available at the timepoint were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 326 | 327
Score on a Scale
  Week 4: number analyzed (Participants) | 325 | 325
  Week 4 | 2.1 (14.17) | 2.2 (13.99)
  Week 12: number analyzed (Participants) | 325 | 325
  Week 12 | 4.9 (16.41) | 1.4 (16.38)
  Week 16 | 5.5 (15.98) | 1.5 (15.78)

56. Secondary Outcome: Change From Baseline in the 36-item Short Form (SF-36) Emotional Problems Subcomponent Score up to Week 16
Description: SF-36 is a generic 36-item questionnaire measuring health-related quality of life. The emotional problem subcomponent is one of the 4 subscales of MCS. The emotional problem subcomponent scores will be calculated by taking a weighted linear combination of the individual question. The score ranges from 0 to 100, with higher values indication poor quality of life. Change from baseline is defined as value at post-baseline visit. A negative change from baseline in SF-36 emotional problems subcomponent indicates an improvement.
Time Frame: Baseline and Week 4, 12 and 16
Population: Randomized population. Only participants with data available at the timepoint were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 326 | 327
Score on a Scale
  Week 4: number analyzed (Participants) | 325 | 325
  Week 4 | 2.718 (20.1133) | 2.128 (20.1154)
  Week 12: number analyzed (Participants) | 325 | 325
  Week 12 | 5.846 (21.4070) | 0.718 (21.0925)
  Week 16 | 7.438 (22.6517) | 2.370 (21.4931)

57. Secondary Outcome: Change From Baseline in the Work Productivity and Activity Impairment (WPAI) Subcomponents Score at Week 16
Description: WPAI contains 4 subcomponents - absenteeism (work time missed), presenteeism (impairment at work/reduced on-the-job effectiveness), work productivity (overall work impairment/absenteeism plus presenteeism), and activity impairment. Each subcomponent score ranges from 0 to 100, with higher numbers indicating worse outcome. Change from baseline is defined as value at post-baseline visit. A negative change from baseline indicates an improvement.
Time Frame: Baseline and week 16
Population: Randomized population. Only participants with data available at the timepoint were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 325 | 325
Score on a Scale
  WPAI Absenteeism: number analyzed (Participants) | 167 | 157
  WPAI Absenteeism | -3.30 (20.777) | 1.23 (19.389)
  WPAI Presenteeism: number analyzed (Participants) | 157 | 149
  WPAI Presenteeism | -13.76 (23.299) | -6.91 (20.332)
  Work Productivity: number analyzed (Participants) | 157 | 149
  Work Productivity | -13.33 (24.053) | -6.80 (21.526)
  WPAI Activity Impairment | -15.20 (25.466) | -9.69 (23.855)

58. Secondary Outcome: Change From Baseline in the European Quality of Life 5D-5L (EQ-5D-5L) Utility Scores and Its Subcomponents up to 16
Description: The European Quality of Life 5D-5L Scale (EQ-5D-5L) assesses general health-related quality of life. Health is defined in 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. Responses are coded so that a '1' indicates no problem, and '5' indicates the most serious problem. The responses for the 5 dimensions are combined in a 5-digit number. Change from Baseline in 5-level EuroQol 5-dimension (EQ-5D-5L) Utility Scores. Change from baseline is defined as value at post-baseline visit. A negative change from baseline indicates an improvement.
Time Frame: Baseline and week 4 and 16
Population: Randomized population. Only participants with data available at the timepoint were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 325 | 325
Score on a Scale
  Utility Score (Week 4) | 0.1006 (0.19470) | 0.0694 (0.19282)
  Utility Score (Week 16) | 0.1630 (0.23696) | 0.0721 (0.23083)
  Mobility (Week 4) | -0.3 (0.77) | -0.3 (0.80)
  Mobility (Week 16) | -0.5 (0.88) | -0.3 (0.92)
  Self-Care (Week 4) | -0.3 (0.81) | -0.2 (0.78)
  Self-Care (Week 16) | -0.5 (0.90) | -0.1 (0.86)
  Usual Activities (Week 4) | -0.3 (0.83) | -0.3 (0.71)
  Usual Activities (Week 16) | -0.5 (0.92) | -0.3 (0.78)
  Pain/Discomfort (Week 4) | -0.4 (0.77) | -0.3 (0.81)
  Pain/Discomfort (Week 16) | -0.6 (0.93) | -0.3 (0.92)
  Anxiety/Depression (Week 4) | -0.2 (0.74) | -0.1 (0.79)
  Anxiety/Depression (Week 16) | -0.3 (0.84) | -0.1 (0.91)

59. Secondary Outcome: Change From Baseline in Patient-Reported Outcome Measures Information System (PROMIS) Sleep Disturbance up to Week 16
Description: The Patient-Reported Outcome Measures Information System Sleep Disturbance assess self-reported perceptions of sleep quality, sleep depth, and restoration associated with sleep. This includes perceived difficulties and concerns with getting to sleep or staying asleep, as well as perceptions of the adequacy of and satisfaction with sleep. The items are evaluated on a 5-point Likert scale ranging from 1 = "not at all" to 5 = "very much" with a 7-day recall period. Higher score means more active disease. Change from baseline is defined as value at post-baseline visit. A negative change from baseline indicates an improvement.
Time Frame: Baseline and week 4, 12, and 16
Population: Randomized population. Only participants with data available at the timepoint were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo
Number analyzed (Participants) | 326 | 326
Score on a Scale
  Week 4: number analyzed (Participants) | 325 | 325
  Week 4 | -1.48 (6.489) | -1.09 (6.413)
  Week 12: number analyzed (Participants) | 325 | 325
  Week 12 | -2.46 (8.196) | -0.88 (8.177)
  Week 16 | -3.15 (7.761) | -1.59 (7.645)

ADVERSE EVENTS:
Time Frame: All-cause mortality and Adverse events were collected from first dose (Day 1) and up to 30 days after the last dose of treatment in the study (up to approximately 164 weeks)
Description: All-cause mortality was collected for all the randomized participants and adverse events were collected for all the treated participants.
Arm/Group | Placebo-Controlled Period - Deucravacitinib 6 mg QD | Placebo-Controlled Period - Placebo | Active Treatment Period - Deucravacitinib 6 mg QD | Active-Treatment Period - Placebo-Deucravacitinib 6 mg QD
All-Cause Mortality (participants affected / at risk) | 0/336 | 0/334 | 0/309 | 0/306
Serious Adverse Events (participants affected / at risk) | 6/332 | 8/333 | 21/309 | 17/306
Other Adverse Events (participants affected / at risk) | 39/332 | 32/333 | 68/309 | 67/306
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo-Controlled Period - Deucravacitinib 6 mg QD (N=332) | Placebo-Controlled Period - Placebo (N=333) | Active Treatment Period - Deucravacitinib 6 mg QD (N=309) | Active-Treatment Period - Placebo-Deucravacitinib 6 mg QD (N=306)
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Sinus node dysfunction (Cardiac disorders) | 0 | 1 | 0 | 0
Iridocyclitis (Eye disorders) | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Alcoholic liver disease (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0 | 0
Hepatitis infectious mononucleosis (Infections and infestations) | 0 | 0 | 0 | 1
Herpes zoster disseminated (Infections and infestations) | 0 | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1
Renal cyst infection (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Vulval cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 1 | 0
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0
Embolic stroke (Nervous system disorders) | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 1
Major depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Vaginal haematoma (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo-Controlled Period - Deucravacitinib 6 mg QD (N=332) | Placebo-Controlled Period - Placebo (N=333) | Active Treatment Period - Deucravacitinib 6 mg QD (N=309) | Active-Treatment Period - Placebo-Deucravacitinib 6 mg QD (N=306)
Nasopharyngitis (Infections and infestations) | 13 | 12 | 24 | 26
Upper respiratory tract infection (Infections and infestations) | 17 | 10 | 32 | 33
Hypertension (Vascular disorders) | 10 | 10 | 18 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-06): https://cdn.clinicaltrials.gov/large-docs/02/NCT04908202/Prot_SAP_000.pdf